CLINICAL TRIAL: NCT03478111
Title: A Randomized, Double-blind, Methotrexate (MTX) Based, Parallel-group, Multicenter Phase III Study to Evaluate Efficacy and Safety of CMAB008 in Adult Patients With Moderately to Severely Active Rheumatoid Arthritis, Compared to Remicade
Brief Title: CMAB008 With MTX Therapy in Adult Patients With Moderately to Severely Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Biomabs Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C008RAIII
Record Dates: First submitted 2018-03-16; First posted 2018-03-27 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAB008+MTX (Experimental): Drug: CMAB008 (recombinant chimeric anti-TNF-α monoclonal antibody injection) infusion of 3mg/kg in Week 0, 2, 6, 14, 22, 30.
  Drug: MIX (methotrexate) will be oral administered at a dose of 7.5mg~15mg weekly from Week 0 to 38.
  Interventions: Drug: CMAB008; Drug: MTX
- Remicade+MTX (Active Comparator): Drug: Remicade (recombinant chimeric anti-TNF-α monoclonal antibody injection) infusion of 3mg/kg in Week 0, 2, 6, 14, 22, 30.
  Drug: MIX (methotrexate) will be oral administered at a dose of 7.5mg~15mg weekly from Week 0 to 38.
  Interventions: Drug: MTX; Drug: Remicade

INTERVENTIONS:
Drug: CMAB008 — the study drug
  Other Names: infliximab
  Arms: CMAB008+MTX
Drug: MTX — basic therapy drug
  Other Names: methotrexate
Drug: Remicade — active comparator
  Other Names: infliximab
  Arms: Remicade+MTX

SUMMARY:
CMAB008 is an infliximab biosimilar candidate. The host cell of Remicade is mouse myeloma SP2/0 cell, however, the host cell of CMAB008 is CHO (Chinese hamster ovary cell). It seems that CMAB008 has lower immunogenicity and higher safety, because Remicade comprises more complex-type and hybrid-type glycans than CMAB008. However, it is not yet known whether CMAB008 is not inferior to Remicade. This randomized, double-blind trial investigates the efficacy and safety of CMAB008 for moderately to severely active rheumatoid arthritis, compared to Remicade.

DETAILED DESCRIPTION:
This is a non-inferiority trial. The primary outcome is the percentage of subjects achieving ACR20. According to the global instruction of Remicade, the effective rate of Remicade is 50%, and the placebo is 20%. Calculate the critical value δ=（50%-20%）×50%=15%, one-side α=0.025, β=0.20, experimental group : control group = 1:1, the results are: CMAB008 group 175 participants, control group 175 participants, 350 participants in total. Take 10% drop-out into consideration, the finial sample sizes are: CMAB008 group 196 participants, control group 196 participants, 392 participants in total.

During the entire duration of the study, all adverse events (AE) and all serious adverse events (SAEs) are collected, fully investigated and documented in source documents and case report forms (CRF). Study duration encompassed the time from when the participant sign the informed consent until the last protocol-specific procedure has been completed, including a safety follow up period.

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the guidelines of Good Clinical Practice (GCP) as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, males or females;
2. Diagnosis of rheumatoid arthritis according to American College of Rheumatology (ACR) 1987 Revised Criteria for the Classification of Rheumatoid Arthritis, and in moderately to severely active stage during screening;
3. Have had one or more DMARDs failure (defined as "failure of traditional/conventional DMARD(s) due to lack of efficacy/desired response or side effects" according to 2015 American College of Rheumatology Guideline for the Treatment of Rheumatoid Arthritis);
4. Non-use of DMARDs (including: Chloroquine, Hydroxychloroquine, Gold Compound, Penicillamine, Salicylazosulfapyridine, Azathioprine, Cyclophosphamide, Cyclosporine A, Leflunomide, Thalidomide etc.) except for MTX in the last 4 weeks before screening;
5. Have completed at least 3 months of treatment with MTX, and steadily at the dosage of 7.5mg~15mg/w at least 4 weeks prior to screening;
6. Non-use of Non-steroidal Anti-inflammatory Drugs (NSAIDs) in the last 2 weeks before enrollment, or if using NSAIDs, should stabilize dose at least 2 weeks;
7. Non-use of glucocorticoid (including intramuscular corticotropin) systematically (e.g., oral administration, intramuscular or intravenous injection) or intra-articular injection; or if concurrent taking glucocorticoid orally, dose (equivalent to the dose of Prednisone) should stabilize≤10mg/d at least 4 weeks;
8. Non-use of Chinese medicine (e.g., Tripterygium, Total Glucosides of Paeony Capsules) for rheumatoid arthritis in the last 4 weeks before screening;
9. Pregnancy test should be negative for procreative female, or not lactating. Both male and female subjects should consent to take effective contraception throughout the study and at least 6 months after the study;
10. Signed the informed consent form;
11. Can participate in visits on schedule;
12. Can understand and complete assessment forms correctly.

Exclusion Criteria:

1. Weight>75Kg;
2. Inoculated live (attenuated) viral/bacterial vaccine in the last 4 weeks before screening;
3. Use of biologicals (including but nor limited to Infliximab, Etanercept, Adalimumab, Tocilizumab, Rituximab etc.) for rheumatoid arthritis in the last 3 months before screening;
4. Severe infection (e.g., acute hepatitis, pneumonia, acute pyelonephritis) in the last 2 months before enrollment, or previous hospitalization due to infection, or previous use of antibiotics, antifungal or antiviral drugs due to infection. However, low-grade infection (e.g., acute upper respiratory infections, simplex urinary tract infection) is not considered as exclusion criteria, whether the subject can be chosen depends on investigator;
5. Suffering from acute infection or recurrent infections disease during screening, e.g., respiratory system infection (influenza, upper respiratory infection, bronchiectasia etc.), acute episode of chronic pyelonephritis, infectious skin wound etc,;
6. Previous opportunistic infection (e.g., herpes zoster, active cytomegalovirus, mycoplasma, pneumocystis pneumonia, histoplasma, aspergillus, mycobacteria except for mycobacterium tuberculosis) in the last 6 months before screening;
7. History of prosthetic joint infections, or suspicious prosthetic joint infections with antibiotic therapy and unremoved prosthetic joint;
8. History of severe hepatic diseases; or HbsAg positive; or only HbcAb positive in Second Liver 5 Indexes, and HBV-DNA positive; or HCV-infected patient;
9. AIDS-infected patient or HIVpositive;
10. One of the following situations relating to tuberculosis:

    1. Concurrent or previous active tuberculosis. Chest X-ray examination (suggest chest anteroposterior and lateral position films) should be performed in the last 3 months before screening, to provide evidence for concurrent or previous tuberculosis;
    2. Intimate contact with active tuberculosis patient recently; or high-risk and/or immunocompromised group (e.g., long-term use of glucocorticoids, immunosuppressor), and with any signs of latent tuberculosis infection;
    3. PPD test (inject 5IU TB-PPD intradermally, measure the diameter of skin induration 72 hours later) performed in the last 3 weeks before screening: diameter of induration≤15mm, and with vesicle or necrosis; or diameter of induration>15mm;
    4. If cannot perform PPD test, perform T-SPOT test: T-SPOT test positive, chest file and clinical evidence indicate that the patient is unsuitable for participation;
11. History of organ allograft operation (except for keratoplasty more than 3 months before the first use of investigational drug);
12. Concurrent or previous malignant tumor (except for total excision and no recurrence of cutaneous squamous cell carcinoma, basal-cell carcinoma or carcinoma in situ of cervix) in the last 5 years before screening;
13. History of lymphoid malignancies (lymphoma) or lymphoproliferative disease; or symptoms and signs indicate that may be lymphoproliferative disease (e.g., lymph node enlargement at neck, clavicle or axilla) during screening; or splenomegaly (≥subcostal 2cm);
14. Concurrent or previous demyelinating diseases of the central nervous system (e.g., multiple sclerosis);
15. Concurrent or previous congestive heart failure;
16. Concurrent or previous other autoimmune disease, and may be expected to affect the assessment of investigational drug;
17. Severe, progressive, uncontrolled cardiovascular, hepatic, renal, pulmonic, gastrointestinal, hematopoietic, endocrine, neural diseases, or other situations that the patient is considered as unsuitable for participation by investigator;
18. History of severe drug or alcohol abuse with clinical symptoms; history of poor drug compliance; or other situations that may interfere protocol compliance (e.g., mental disease, frequent travel, lack of willingness);
19. Laboratory tests results meet one of the following indexes: HGB<8.5g/dL, WBC<3.5*10^9/L, PLT<80*10^9/L, ALT/AST>2*upper limit of normal value, CREA>upper limit of normal value;
20. Allergic reaction against human immunoglobulin, infliximab or other ingredient;
21. Participation in another drug clinical trial in the last 30 days before screening or within 5 half-lives of drug (longer time shall prevail).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects achieving ACR20 | Baseline up to 30 weeks
  Defined as the percentage of subjects achieving ACR20 of all subjects

SECONDARY OUTCOMES:
The percentage of subjects achieving ACR20 | Baseline up to 2,6,14,22 weeks
  Defined as the percentage of subjects achieving ACR20 of all subjects
The percentage of subjects achieving ACR50,70 | Baseline up to 2,6,14,22,30 weeks
  Defined as the percentage of subjects achieving ACR50,70 of all subjects
Improvement rate of the duration of morning stiffness | Baseline up to 2,6,14,22,30 weeks
  Improvement rate=(before the treatment - after the treatment)/before the treatment *100%
Improvement rate of the number of joint swelling or tenderness | Baseline up to 2,6,14,22,30 weeks
  Improvement rate=(before the treatment - after the treatment)/before the treatment *100%
Improvement rate of Visual Analogue Scale (VAS) | Baseline up to 2,6,14,22,30 weeks
  Improvement rate=(before the treatment - after the treatment)/before the treatment *100%.
  Visual Analogue Scale(VAS) is designed to present to the respondent a rating scale. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced. VAS data of this type is recorded as the number of centimeters from the left of the line with the range 0-10.
  No pain <-- 10 cm. --> Pain as bad as possible
Improvement rate of Health Assessment Questionnaire (HAQ) score | Baseline up to 2,6,14,22,30 weeks
  Improvement rate=(before the treatment - after the treatment)/before the treatment *100%.
  The Health Assessment Questionnaire (HAQ) Disability Index assesses a patient's level of functional ability. There are 20 questions in eight categories of functioning which represent a comprehensive set of functional activities - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. The patient's responses are made on a scale from zero (no disability) to three (completely disabled).
Improvement rate of physicochemical indexes of curative effect (ESR, CRP) | Baseline up to 2,6,14,22,30 weeks
  Improvement rate=(before the treatment - after the treatment)/before the treatment *100%

CONTACTS AND LOCATIONS:
Overall Officials: Yin Su, Ph.D, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye H, Liu S, Xu J, Chai K, He D, Fang Y, Xie Q, Liu H, Liu Y, Hua B, Hu J, Zhang Z, Zhou M, Zhao D, Li Y, Jiang Z, Wang M, Li J, Zhang Z, Li X, Li Y, Sun E, Bi L, Wei W, Tie N, He L, Huang X, Zhang Y, Huang Q, Wang X, Liu X, Li J, Su Y. Efficacy and Safety of CMAB008 Compared with Innovator Infliximab in Patients with Moderate-to-Severe Rheumatoid Arthritis Receiving Concomitant Methotrexate: A Randomized, Double-blind, Multi-center, Phase III Non-inferiority Study. Rheumatol Ther. 2023 Jun;10(3):757-773. doi: 10.1007/s40744-023-00544-2. Epub 2023 Mar 25. PMID 36964872
- [Derived] Su Y, Li J, Wang C, Zhang X, Hou S, Guo H, Deng C, Ou L, Wang J. Population Pharmacokinetics of CMAB008 (an Infliximab Biosimilar) and Remicade(R) in Healthy Subjects and Patients with Moderately to Severely Active Rheumatoid Arthritis. Adv Ther. 2023 Mar;40(3):1005-1018. doi: 10.1007/s12325-022-02396-8. Epub 2023 Jan 6. PMID 36607544